CLINICAL TRIAL: NCT06564311
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Obexelimab in Patients With Relapsing Multiple Sclerosis
Brief Title: A Study of Obexelimab in Patients With Relapsing Multiple Sclerosis (MoonStone)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zenas BioPharma (USA), LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZB012-02-002
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-06

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Relapsing Multiple Sclerosis; RMS; MS; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: This is a Phase 2, multicenter, double-blind, placebo-controlled study to evaluate the efficacy and safety of obexelimab in patients with RMS. The study consists of a Screening Period (Day 28 to Day -1), followed by a 24-week Treatment Period (Part A or RCP consists of 12 doses of obexelimab or placebo; Part B or OLP consists of 12 doses of open-label obexelimab), a 52-week OLE and an expected 12-week Follow-up Period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, Care Providers, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obexelimab (Experimental): Obexelimab will be administered as a subcutaneous injection for 76 weeks
  Interventions: Drug: Obexelimab
- Placebo (Placebo Comparator): Placebo will be administered as a subcutaneous injection for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Obexelimab — Obexelimab is a monoclonal antibody that simultaneously binds CD19 and FcyRIIb, resulting in down regulation of B cell activity
  Arms: Obexelimab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study aims to examine the efficacy and safety of obexelimab in participants with relapsing multiple sclerosis

DETAILED DESCRIPTION:
The study consists of a Screening Period (Day -28 to Day -1), a 24-week treatment period (Part A and Part B), a 52 week open label extension and an expected 12-week Follow-up Period. Patients with Relapsing Multiple Sclerosis will be randomized in 2:1 ratio to obexelimab or placebo. Randomization will be stratified by Gd lesion status at screening (≥ 1 vs 0).

Part A is the 12-week Randomized Placebo-Controlled Period (RCP), during which obexelimab or placebo will be administered as weekly subcutaneous (SC) injections. Following Part A, all patients will enter the Part B, a 12-week Open-Label Period (OLP), during which all patients will receive obexelimab administered as weekly SC injections. After Part B, patients will enter Part C, a 52-week Open-Label Extension (OLE), after which they will return for an in-clinic Safety Follow-Up Visit 12 weeks after the completion of Part C (i.e. Week 88). If at this time, B cells have not returned to baseline or above the lower limit of normal (LLN), patients will be asked to return every 12 weeks until B cells return to baseline or above the LLN (at minimum). The maximum expected duration of the study is 92 weeks (Screening Period = 4 weeks, Parts A, B and C = 76 weeks, Follow-up Period = 12 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of RMS (relapsing-remitting or secondary progressive with relapses) according to the 2017 revision of the McDonald diagnostic criteria
2. An EDSS of ≤ 5.5 at the Screening Visit
3. Must have documentation of:

   1. . at least 1 relapse within the previous year OR
   2. . ≥ 2 relapses within the past 2 years OR
   3. . ≥ 1 active Gd-enhancing brain lesion on an MRI scan within the past 6 months prior to screening
4. Not of childbearing potential or willing to follow contraceptive guidance

Exclusion Criteria:

1. Primary progressive MS or secondary progressive MS without relapses
2. Meet criteria for neuromyelitis optica spectrum disorder
3. Relapse in the 30 days prior to randomization
4. ≥ 10 years disease duration from onset with patient's EDSS ≤ 2.0 (patient reported is adequate in absence of written medical record)
5. Has > 20 Gd+ lesions on brain MRI at screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Cumulative number of new GdE T1 hyperintense lesions | Week 8 and Week 12
  Cumulative number of new GdE T1 hyperintense lesions as measured by brain MRI

SECONDARY OUTCOMES:
Number of T2 Lesions | Week 8 and Week 12
  cumulative number of new and/or enlarging T2 weighted hyperintense lesions
Number of GdE T1 lesions | Week 4, Week 8, and Week 12
  number of new GdE T1 hyperintense lesions
Volume of T2 lesions | Week 12
  change from baseline in volume of T2 lesions
Serum NfL | Week 12
  serum NfL
Incidence of Adverse Events, injection site reactions and hypersensitivity reactions | 24 weeks
  Incidence of Adverse Events, injection site reactions and hypersensitivity reactions, serious adverse events, and adverse events of special interest, as defined by the CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (47):
- United States (14):
  - North Central Neurology, Cullman, Alabama
  - Center for Neurology and Spine, Phoenix, Arizona
  - Perseverance Research Center, Scottsdale, Arizona
  - Regina Berkovich MD PhD, Inc, West Hollywood, California
  - Aqualine Clinical Research, Naples, Florida
  - University of South Florida, Tampa, Florida
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Infusion Associates Plymouth, Plymouth, Minnesota
  - MS Center for Innovations in Care, St Louis, Missouri
  - Holy Name Medical Center, Teaneck, New Jersey
  - Boster Center for MS, Columbus, Ohio
  - North Texas Institute of Neurology and Headache, Plano, Texas
  - Center for Neurological Disorders, Greenfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Neuro-logisch Wien, Vienna, Austria
- Belgium (2):
  - Rehabilitation & MS Center, Noorderhart Hospital, Overpelt
  - AZ Delta-Deltalaan 1, Roeselare
- China (5):
  - Tiantan Hospital, Capital Medical University, Beijing
  - The First Affiliation Hospital of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - People's Hospital of Xinjiang Uyaur Autonomous Region, Ürümqi
  - Tongji Hospital, Tongji Medical Center of HUST, Wuhan
- Klinicki bolnicki centar Zagreb, Zagreb, Croatia
- Czechia (3):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Nemocnice Jihlava, Jihlava
  - General University Hospital Praha, Prague
- Aalborg Universitetshospital, Aalborg, Denmark
- Greece (2):
  - Attikon University General Hospital, Chaïdári
  - University General Hospital of Larissa, Larissa
- Italy (4):
  - Fondazione Isituto G. Giglio di Cefalu, Cefalù
  - University of Florence, Florence
  - Istituto Neurologico Mediterraneo Neuromed, Pozzilli
  - Fondazione PTV Policlinico Tor Vergata, Roma
- Poland (4):
  - Neurocentrum Bydgoszcz sp.z o.o., Bydgoszcz
  - M.A. LEK A.M. Maciejowsy Spolka Cywilna, Katowice
  - Zanamed Medical Clinic Sp z o.o., Lublin
  - Wielospecjalistyczne Centrum Medyczne Ibismed, Zabrze
- Spain (7):
  - Hospital Clinico San Carlos, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen de La Arrixaca, Murcia
  - Hospital Virgen Macarena, Seville
  - Hospipal La Fe Valencia, Valencia
- United Kingdom (3):
  - Leicester General Hospital, Leicester
  - Barts Health NHS Trust, London
  - Morriston Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Undecided